CLINICAL TRIAL: NCT06366360
Title: Rehabilitation of Unilateral Spatial Neglect Using an Immersive Virtual Reality Music Practice Program
Brief Title: Immersive Virtual Reality Treatment for Unilateral Spatial Neglect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Principal Investigator, Silvia Silvestri, Medical Doctor, Hopitaux de Saint-Maurice
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Piano-Neglect
Record Dates: First submitted 2024-03-27; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Unilateral Spatial Neglect
Keywords: Rehabilitation; Unilateral Spatial Neglect; Immersive Virtual Reality; Music
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Each patient was assigned to a group that received 2 rehabilitations for 4 weeks, 1) both Immersive virtual reality therapy and a conventional rehabilitation first, and then conventional rehabilitation alone, or 2) A conventional rehabilitation alone and then both Immersive virtual reality therapy, and conventional rehabilitation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality rehabilitation first (Active Comparator): Each patient received 2 rehabilitations: both an immersive virtual reality and a conventional rehabilitation first (during 2 weeks), and then conventional rehabilitation alone (during 2 weeks)
  Interventions: Other: Immersive Virtual Reality Intervention; Other: Conventional rehabilitation
- Conventional rehabilitation first (Active Comparator): Each patient received 2 rehabilitations: a conventional rehabilitation alone first (during 2 weeks), and then both conventional rehabilitation and immersive virtual reality rehabilitation (during 2 weeks)
  Interventions: Other: Immersive Virtual Reality Intervention; Other: Conventional rehabilitation

INTERVENTIONS:
Other: Immersive Virtual Reality Intervention — The immersive virtual reality rehabilitation protocol is an experimental protocol based on musical practice. This protocol will be based on the "Piano Vision" application, which allows several modes of music production: free or guided musical practice.
Other: Conventional rehabilitation — The conventional rehabilitation corresponds to the classically performed in the cognitive treatment of unilateral spatial neglect. It involves training visual scanning using barrage exercises, sequence identification, scene description, and pointing.

SUMMARY:
Unilateral Spatial Neglect (USN) is a relatively common neuropsychological syndrome following stroke. It is characterized by difficulties in detecting, orienting and identifying events located in the hemispace contralateral to a brain lesion, unrelated to a primary motor or sensory disorder. Numerous methods have been developed for the rehabilitation of this syndrome. However, limitations in terms of efficacy are highlighted. These limitations may be linked to the fact that these methods are restricted to certain sensory modalities, thus failing to take into account the heterogeneity of the syndrome. Moreover, some patients' adherence to rehabilitation programs can also be complicated by motivational difficulties. Immersive Virtual Reality could help overcome these limitations. Indeed, it enables the introduction of new sensory modalities, notably auditory, to support a better apprehension of space.

The main objective of this study is to determine the efficacy of an immersive virtual reality rehabilitation protocol based on musical practice in patients suffering from USN. This study also aims to explore the benefits of this rehabilitation protocol on patients' daily lives, as well as to explore the influence of patients' mood and motivation on the benefits of the immersive virtual reality rehabilitation protocol.

To achieve these goals, patients will benefit from immersive virtual reality rehabilitation based on music practice. This rehabilitation will be compared to conventional USN rehabilitation. To this end, patients will be divided into two groups: classical rehabilitation only or classical rehabilitation and immersive virtual reality in parallel. Each patient will be randomly assigned to one of the two groups for a period of 2 weeks. Pre- and post-rehabilitation assessments will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Free and informed written consent
* Enrolled in the French social security system
* Cerebral lesion of vascular origin
* Unilateral spatial neglect syndrome

Exclusion Criteria:

* Epilepsy or migraine
* Major vision problems
* Major hearing impairment
* Pre-existing cognitive impairment (MMSE < 20)
* Major disorders of verbal comprehension preventing the protocol
* Refusal to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Bells Test | 8 weeks
  The patient has to circle 35 bells placed on an A4 sheet between distractors. The number of total and lateralized omissions is examined. The minimum value corresponds to the absence of omissions and the maximum value corresponds to the total number of stimuli (35 bells) or the number of lateralized stimuli (15 bells in each hemifield). Specifically, if the total number of omissions is greater than 6, or the difference in omissions between the two sides of the sheet is greater than 2, the patient is considered deficient.
Mesulam cancellation Task | 8 weeks
  The patient has to cross out a target stimulus (the letter A) among other distracting letters arranged on a sheet of A4 paper.
  The number of total and lateralized omissions on each side of the sheet is analyzed. A maximum score of 60 omissions can be recorded. 30 lateralized omissions is possible and a minimum score of 0 lateralized omissions is also possible.
Bisection Test | 8 weeks
  The patient must cut the lines of different lengths (20 cm and 5 cm) into two equal parts.
  The minimum value corresponds to a bisection at the center of the stimuli and the maximum value corresponds to a bisection at the contralesional end of this stimulus. More specifically, for the 20 cm lines, a deviation of +6.5 mm or -7.3 mm is considered a deficit, and for the 5 cm lines, a deviation of +2 mm or -2 mm is considered a deficit.
Copying Test | 8 weeks
  The patient has to copy a figure representing a house with trees on both sides on a sheet of A4 paper.
  Each element of the drawing is individually marked with a score of 0 (if not represented or poorly represented) or 1 (if well represented). The omission of an element is considered a deficit and corresponds to a score below the maximum of 6.
Scene description Task | 8 weeks
  The patient has to describe the objects in a visual scene presented on an A3 sheet of paper and placed in front of him or her.
  The number of omissions in each part of the picture is analyzed. The total score is between 0 and 3: 0 corresponds to 3 or more omissions, 1 to 2 omissions, 2 to 1 omission, and 3 to no omissions. The patient is considered to be deficient if the score exceeds 0.
Ecological scale of daily life activities | 8 weeks
  The patient and a therapist or family member complete a scale that asks questions about everyday activities.
  The patient must answer 10 questions, each of which is scored from 0 to 3 according to the severity criterion. 0 corresponds to no neglect and 3 to significant neglect, so the minimum score is 0 and the maximum is 30. If a patient receives a score equal to or greater than 1, he is considered neglected.
Piano bisection Task | 8 weeks
  The patient must indicate which key corresponds to the middle key of the piano. It's a qualitative measure. There are no minimum or maximum values among the 61 piano keys. However, the investigators can consider the minimum to be the actual center key of the piano and the maximum to be the contralesional key of the piano.
Identifying the keys at the ends of the piano | 8 weeks
  The patient must indicate which keys are furthest to the left and right of the piano.
  It's a qualitative measure. The maximum value can be considered as the touch at the contralesional end, and the minimum as the touch at the ipsilesional end.
Virtual reality Bells Test | 8 weeks
  The patient is asked to perform the same task as in the classical test, but this time the bells are placed in a virtual environment 120° around the patient.
  As in the classical version, the number of total and lateralized omissions is assessed. The minimum value corresponds to the absence of omissions and the maximum value corresponds to the total number of stimuli (35 bells) or the number of lateralized stimuli (15 bells in each hemifield).
Auditory Stimuli Localization Task in virtual reality | 8 weeks
  The patient must localize auditory stimuli in a 180° horizontal virtual environment to a precise point in the virtual environment.
  The difference between the real position of the sound and the position targeted by the patient is examined. The minimum value corresponds to no difference and the maximum value corresponds to a maximum difference between these two coordinates.
Ecological virtual reality bisection task | 8 weeks
  The patient has to cut bread sticks of different size into 2 equal parts. The minimum value corresponds to a bisection at the center of the stimulus and the maximum value corresponds to a bisection at the contralesional end of this stimulus. For each stimulus, a calculation is made between the value reported by the patient and the actual expected value.
Virtual reality Baking Tray test | 8 weeks
  The patient must place 16 pieces of dough evenly on a baking tray. The minimum value corresponds to an equal distribution between the 2 hemispaces of the tray (i.e. 8 pieces of dough on each side) and the maximum value corresponds to the positioning of all pieces in the contralesional hemispace. A difference of more than 2 cubes indicates a deficit.

SECONDARY OUTCOMES:
Mood assessment | 4 weeks
  At the beginning and end of each session, patients are asked to rate their mood on a visual analog scale from 1 to 10 to quantify the impact of their mood on the treatment.
Situational motivation questionnaire | 4 weeks
  Before and after each intervention, patients are asked to complete a Situational Motivation Questionnaire to assess the impact of their words on their health.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux de Saint-Maurice, Saint-Maurice, France